CLINICAL TRIAL: NCT03929250
Title: A Pharmacokinetic Study of Centella Asiatica in the Elderly
Brief Title: Pharmacokinetics of Centella Asiatica in the Elderly
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amala Soumyanath, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00017697
Record Dates: First submitted 2019-04-21; First posted 2019-04-26 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Elderly

STUDY DESIGN:
Intervention Model Description: Randomization will use an arm equivalence design to promote equal numbers of participants for each order schema.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2g CAW Dose, then 4g CAW Dose (Experimental): Participants first receive a single dose of a product containing 2g CAW, then after a minimum washout period of 2 weeks, they receive a single dose of a product containing 4g CAW.
  Interventions: Drug: 2g Centella asiatica water extract product; Drug: 4g Centella asiatica water extract product
- 4g CAW Dose, then 2g CAW Dose (Experimental): Participants first receive a single dose of a product containing 4g CAW, then after a minimum washout period of 2 weeks, they receive a single dose of a product containing 2g CAW.
  Interventions: Drug: 2g Centella asiatica water extract product; Drug: 4g Centella asiatica water extract product

INTERVENTIONS:
Drug: 2g Centella asiatica water extract product — 2g Centella asiatica water extract product is a powder containing Centella asiatica water extract (CAW) and excipients to improve palatability, color matching and dispersability in water. It will be consumed on an empty stomach orally suspended in 10-12 ounces of water.
  Other Names: CAP 2g
Drug: 4g Centella asiatica water extract product — 4g Centella asiatica water extract product is a powder containing Centella asiatica water extract (CAW) and excipients to improve palatability, color matching and dispersability in water. It will be consumed on an empty stomach orally suspended in 10-12 ounces of water.
  Other Names: CAP 4g

SUMMARY:
This study will measure the oral bioavailability and pharmacokinetics of known bioactive compounds from a standardized Centella asiatica water extract (CAW) product (CAP) in cognitively healthy elders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To assess the bioavailability and rate of clearance of Centella asiatica derived compounds in the plasma and urine of cognitively healthy elders over 12 hours.
2. To determine the acute tolerability of a Centella asiatica product in cognitively healthy elders.

OUTLINE:

Participants will orally consume a single administration of a standardized Centella asiatica water extract product (CAP). Two doses (2g and 4g CAW) will be administered on separate occasions, at least two weeks apart. The levels of known bioactive compounds present in Centella asiatica will be measured in human plasma and urine over 12 hours after administration of each of the doses.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65-85, male and female
2. Sufficient English language skills to complete all tests
3. Sufficient vision and hearing to complete all tests
4. No known allergies to Centella asiatica or CAP components
5. Willingness to discontinue all botanical dietary supplements for one week prior to and during each study visit
6. Willingness to comply with a 48-hour low plant diet for each study visit
7. Absence of significant depression symptoms (Geriatric Depression Scale-15 score of <12)
8. Body Mass Index (BMI) greater than 17 and less than 35 at screening
9. Non-demented, defined as Clinical Dementia Rating (CDR) score of zero and Mini Mental State Examination (MMSE) score >28
10. General health status that will not interfere with the ability to complete the study

Exclusion Criteria:

1. Current smoking, alcohol or substance abuse according to DSM-V criteria
2. Women who are pregnant, planning to become pregnant or breastfeeding
3. Men who are actively trying to conceive a child or planning to within three months of study completion
4. Severe aversion to venipuncture
5. Abnormal laboratory evaluation indicating asymptomatic and untreated urinary tract infection
6. Cancer within the last five years, with the exception of localized prostate cancer (Gleason Grade <3) and non-metastatic skin cancers
7. Comorbid conditions such as diabetes mellitus, kidney failure, liver failure, hepatitis, blood disorders, clinical symptomatic orthostatic hypotension, and unstable or significantly symptomatic cardiovascular disease
8. Significant disease of the central nervous system such as brain tumor, seizure disorder, subdural hematoma, cranial arteritis, or clinically significant stroke
9. Major depression, schizophrenia, or other major psychiatric disorder defined by DSM-V criteria
10. Medications: sedatives (except those used occasionally for sleep), central nervous system active medications that have not been stable for two months (including beta blockers, cimetidine, SSRIs, SNRIs), anticoagulants (i.e. Warfarin), investigational drugs used within five half-lives of baseline visit, systemic corticosteroids, neuroleptics, anti-Parkinsonian agents, narcotic analgesics, nicotine (tobacco, patches, gum, lozenges, etc.), Cannabis sativa (herb or edibles)
11. Diseases associated with dementia such as Alzheimer's disease, vascular dementia, normal pressure hydrocephalus or Parkinson's disease with a CDR score >0.5 and MMSE score <28
12. Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amala Soumyanath, PhD, Principal Investigator — OHSU Department of Neurology
Locations (1):
- Oregon Health and Science University Department of Neurology, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results reported in a publication after de-identification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Immediately after publication and for a period of 3 years following publication.
Access Criteria: Anyone who wishes access to the data, for any reason. Requests should be directed to Dr Amala Soumyanath at soumyana@ohsu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- 2g CAW Dose, Then 4g CAW Dose: Participants first receive a single dose of product containing 2g CAW, then after a minimum washout period of 2 weeks, they receive a single dose of product containing 4g CAW.
- 4g CAW Dose, Then 2g CAW Dose: Participants first receive a single dose of product containing 4g CAW, then after a minimum washout period of 2 weeks, they receive a single dose of product containing 2g CAW.
Period: Overall Study
Arm/Group | 2g CAW Dose, Then 4g CAW Dose | 4g CAW Dose, Then 2g CAW Dose
Started | 4 | 4
Completed | 4 | 3
Not Completed | 0 | 1
Not completed — Blood draws could not be successfully obtained | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants including those in the (a) 2g CAW, then 4g CAW arm or (b) 4g CAW then 2g CAW arm
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (1.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 125 (4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 78 (2)
Body temperature [Mean (Standard Deviation); unit: degrees Fahrenheit] | 98.3 (0.2)
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 67 (4)
White blood cell [Mean (Standard Deviation); unit: 10^3 cells/cu mm] | 6.7 (0.4)
Red blood cell [Mean (Standard Deviation); unit: 10^6 cells/cu mm] | 5.0 (0.2)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 15.3 (0.5)
Hematocrit [Mean (Standard Deviation); unit: percentage] | 46.4 (1.4)
Platelet [Mean (Standard Deviation); unit: 10^3 cells/cu mm] | 233.9 (7.5)
Blood glucose [Mean (Standard Deviation); unit: mg/dL] | 90.6 (4.3)
Blood urea nitrogen [Mean (Standard Deviation); unit: mg/dL] | 15.8 (1)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.6)
total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.5 (0.03)
Aspartate aminotransferase [Mean (Standard Deviation); unit: U/L] | 24.6 (0.7)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 30.1 (2.5)
Total protein [Mean (Standard Deviation); unit: g/dL] | 7.4 (0.1)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.0 (0.1)
Sodium [Mean (Standard Deviation); unit: mmol/L] | 140.5 (0.5)
Chloride [Mean (Standard Deviation); unit: mmol/L] | 106.5 (0.5)
Potassium [Mean (Standard Deviation); unit: mmol/L] | 4.0 (0.1)
Total CO2 [Mean (Standard Deviation); unit: mmol/L] | 28.9 (0.5)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 9.2 (0.1)
Anion gap [Mean (Standard Deviation); unit: mEq/L] | 5.3 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Human Plasma Concentration of Bioactives From Centella Asiatica.
Description: Following oral administration of a product made from a water extract of Centella asiatica (CAP), the plasma concentration of Centella asiatica derived bioactive compounds (triterpenes, caffeoylquinic acids, and their metabolites) will be measured in blood samples obtained over a 12 hour period, using high performance liquid chromatography tandem mass spectrometry in order to generate a pharmacokinetic curve, and determine pharmacokinetic parameters (maximum concentration and area under the curve) for each of the two doses (2g and 4g).
Time Frame: A 12-hour post-administration period (15, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, and 720 minutes).
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- 2g CAW Dose: 2g of Centella asiatica water extract in a standardized product.
  2g Centella asiatica water extract product: 2g Centella asiatica water extract product is a powder containing Centella asiatica water extract and excipients to improve palatability, color matching and dispersability in water. It will be consumed on an empty stomach orally suspended in 10-12 ounces of water.
- 4g CAW Dose: 4g of Centella asiatica water extract in a standardized product.
  4g Centella asiatica water extract product: 4g Centella asiatica water extract product is a powder containing Centella asiatica water extract and excipients to improve palatability, color matching and dispersability in water. It will be consumed on an empty stomach orally suspended in 10-12 ounces of water.
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
ng/mL
  Asiatic acid | 174 (22) | 372 (53)
  Caffeic acid | 0.3 (0.1) | 0.5 (0.1)
  Dihydrocaffeic acid | 0.4 (0.1) | 0.5 (0.1)
  Dihydroferulic acid | 9.3 (4.4) | 8.1 (2.9)
  Dicaffeoylquinic acids | 1.2 (0.6) | 1.9 (0.8)
  Ferulic acid | 1.5 (0.3) | 1.5 (0.6)
  3-(3-hydroxyphenyl)propionic acid | 5.8 (3.0) | 10.6 (2.9)
  Isoferulic acid | 1.5 (0.8) | 1.5 (0.4)
  Madecassic acid | 107 (18) | 197 (43)
  Monocaffeoylquinic acids | 1.6 (0.5) | 4.2 (1.4)

2. Primary Outcome: Total Plasma Concentration Over Time (Area Under the Curve) From Centella Asiatica Water Extract Product.
Description: as for outcome 1
Time Frame: A 12-hour post-administration period (15, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, and 720 minutes).
Measure: Mean (Standard Error); unit: ng/mL*hr
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
ng/mL*hr
  Asiatic acid | 48755 (7152) | 91330 (17723)
  Caffeic acid | 1.8 (0.5) | 2.4 (0.6)
  Dihydrocaffeic acid | 1.7 (0.6) | 1.9 (0.5)
  Dihydroferulic acid | 35.6 (18.6) | 41.0 (12.7)
  Dicaffeoylquinic acids | 3.4 (1.8) | 5.0 (1.5)
  Ferulic acid | 11.3 (2.9) | 9.9 (2.8)
  3-(3-hydroxyphenyl)propionic acid | 56.8 (31.7) | 50.2 (15.1)
  Isoferulic acid | 5.3 (1.6) | 7.4 (1.6)
  Madecassic acid | 26771 (3585) | 48373 (12476)
  Monocaffeoylquinic acids | 6.2 (2.4) | 10.1 (3.9)

3. Primary Outcome: Half-life
Description: The half-life (t1/2) of the known bioactive compounds was calculated from the plasma concentrations measured by high performance liquid chromatography tandem mass spectrometry to help determine dosage intervals.
Time Frame: A 12-hour post-administration period (15, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, and 720 minutes).
Measure: Mean (Standard Error); unit: hours
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
hours
  Asiatic acid | 4.1 (0.7) | 4.9 (1.3)
  Caffeic acid | 8.4 (3) | 10.3 (3.7)
  Dihydrocaffeic acid | 1.8 (1.2) | 1.9 (0.8)
  Dihydroferulic acid | 7.1 (1.7) | 6.6 (3.8)
  Dicaffeoylquinic acids | 2 (1.2) | 2.6 (1.8)
  Ferulic acid | 14.1 (3.9) | 2.9 (1.3)
  3-(3-hydroxyphenyl)propionic acid | 5 (2) | 2.6 (0.5)
  Isoferulic acid | 7 (2.4) | 3.5 (0.5)
  Madecassic acid | 9.2 (3.7) | 6.7 (0.8)
  Monocaffeoylquinic acids | 3.4 (1.1) | 1.7 (1.1)

4. Primary Outcome: Time of Maximum Concentration
Description: The time of maximum concentration (tmax) of the known bioactive compounds and their metabolites will be calculated from the concentrations measured by high performance liquid chromatography tandem mass spectrometry in order to help determine dosage intervals
Time Frame: A 12-hour post-administration period (15, 30, 45, 60, 90, 120, 180, 240, 360, 480, 600, and 720 minutes).
Measure: Mean (Standard Error); unit: hours
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
hours
  Asiatic acid | 2.2 (0.4) | 2.8 (0.2)
  Caffeic acid | 5.3 (1.9) | 4.5 (1.6)
  Dihydrocaffeic acid | 6.1 (1.7) | 3.2 (1.3)
  Dihydroferulic acid | 5.9 (1.6) | 5.7 (1.5)
  Dicaffeoylquinic acids | 3.7 (1.9) | 4.3 (1.7)
  Ferulic acid | 5.9 (1.3) | 7.1 (1.2)
  3-(3-hydroxyphenyl)propionic acid | 7.4 (1.5) | 5.7 (0.7)
  Isoferulic acid | 2.4 (1) | 1 (0.32)
  Madecassic acid | 2.4 (0.3) | 2.7 (0.2)
  Monocaffeoylquinic acids | 1.2 (0.4) | 3.4 (1.2)

5. Secondary Outcome: Urinary Excretion
Description: The concentration of bioactive compounds from Centella asiatica (triterpenes, caffeoylquinic acids, and their metabolites) will be measured in a pooled urine sample collected over 12 hours after CAP administration and analyzed using high performance liquid chromatography tandem mass spectrometry.
Time Frame: Over 12 hours post-administration
Measure: Mean (Standard Error); unit: micrograms
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
micrograms
  Asiatic acid | 0 (0) | 0 (0)
  Asiaticoside | 20.7 (6.7) | 18.6 (4.5)
  Caffeic acid | 42.8 (11.6) | 48.7 (9.3)
  Dihydrocaffeic acid | 26.8 (10) | 24.8 (6.1)
  Dihydroferulic acid | 225.5 (83.5) | 225.1 (94.8)
  Dicaffeoylquinic acids | 0 (0) | 0 (0)
  Ferulic acid | 146.8 (33.5) | 137.4 (24.6)
  3-(3-hydroxyphenyl)propionic acid | 223.4 (76.7) | 247.9 (73.6)
  Isoferulic acid | 65.9 (23.1) | 225.1 (15.9)
  Madecassic acid | 0 (0) | 0 (0)
  Madecassoside | 0 (0) | 0 (0)
  Monocaffeoylquinic acids | 21.3 (8.6) | 19.3 (2.6)

6. Secondary Outcome: Oral Temperature
Description: Oral temperature will be measured in degrees Fahrenheit by means of a thermometer.
Time Frame: 720 minutes after administration
Measure: Mean (Standard Error); unit: degrees Fahrenheit
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
degrees Fahrenheit | 98.2 (0.1) | 98.1 (0.1)

7. Secondary Outcome: Pulse Rate
Description: Pulse rate will be measured peripherally over one minute.
Time Frame: 720 minutes after administration
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
beats per minute | 69 (4) | 64 (3)

8. Secondary Outcome: Seated Systolic Blood Pressure
Description: Seated blood pressure will be measured in millimeters mercury.
Time Frame: 720 minutes after administration
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
mmHg | 125 (4) | 119 (5)

9. Secondary Outcome: Body Mass Index
Description: Height in centimeters and weight in kilograms will be measured and aggregated to measure body mass index in kilograms per meter squared (kg/m2).
Time Frame: 720 minutes after administration
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
kg/m^2 | 28.4 (1.3) | 28 (1.4)

10. Secondary Outcome: Participants With Change in Electrocardiography
Description: Resting electrocardiography will be measured for up to five minutes using a five lead mobile electrocardiogram. The investigators will determine the number of participants who develop changes in electrocardiography compared to the zero minute timepoint following CAP administration.
Time Frame: 0, 360 and 720 minutes after administration
Measure: Count of Participants; unit: Participants
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
Participants | 0 | 0

11. Secondary Outcome: Seated Diastolic Blood Pressure
Description: Seated blood pressure will be measured in millimeters mercury.
Time Frame: 720 minutes after administration
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 2g CAW Dose | 4g CAW Dose
Number analyzed (Participants) | 7 | 8
mmHg | 74 (3) | 69 (1)

ADVERSE EVENTS:
Time Frame: 0, 6, 12 and 24 hours after administration of each dose level (2g CAW or 4g CAW)
Description: A standard multi-system questionnaire will record the type and severity (range 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal) of any adverse events.
Arm/Group | 2g CAW Dose | 4g CAW Dose
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2g CAW Dose (N=8) | 4g CAW Dose (N=8)
Excessive sleep (General disorders) | 1 (1) | 0 (0)
Disappointment (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Boredom (Social circumstances) | 0 (0) | 1 (1)
Weakness/fatigue (General disorders) | 0 (0) | 1 (1)
Musculoskeletal pain or stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Fainting/dizziness (Cardiac disorders) | 3 (3) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral edema or swelling (Vascular disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gas/indigestion (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increased thirst (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal or metallic taste in mouth (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal pain/cramps (Gastrointestinal disorders) | 1 (1) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Increased urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine color change (Renal and urinary disorders) | 1 (1) | 2 (2)
Itchiness/dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin color change (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Redness (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash/hives (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin puffiness/ tissue fluid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis, indurate (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 1 (1)
Weight loss (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03929250/Prot_SAP_000.pdf